CLINICAL TRIAL: NCT06073743
Title: The Effect of Video Based Games Exercise Training on Selective Motor Control, Fear of Falling and Functional Capacity in Individuals With Spastic Cerebral Palsy
Brief Title: Video Based Games Exercise Training in Individuals With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIBU-FTR-ST-03
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Spastic Cerebral Palsy
Keywords: Spastic cerebral palsy; Virtual reality; Selective motor control; Fear of falling; Functional capacity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy Group (Active Comparator): 30 minutes of upper and lower extremity strengthening exercises, upper and lower extremity stretching exercises, functional exercises to increase joint range of motion, tone regulation exercises, 30 minutes of weight transfer exercises to the upper and lower extremities, exercises to improve elective motor control (including isolated joint movements). exercises), balance and coordination exercises (weight transfer to the right-left, front-back on the balance board, cross-arm-leg exercises, exercises for balance and protective reactions), walking training will be applied.
  Interventions: Other: Conventional Physiotherapy
- Video Game Based Exercise Training Group (Experimental): 30 minutes of upper and lower extremity strengthening exercises, upper and lower extremity stretching exercises, functional exercises to increase joint range of motion, tone regulation exercises, 30 minutes of XBox Video Games (10 minutes of Reflex Ridge, 10 minutes of Rallyball, 10 minutes of River rush games) will be applied.
  Interventions: Other: Conventional Physiotherapy; Other: Video Game Based Exercise Training

INTERVENTIONS:
Other: Conventional Physiotherapy — The conventional physiotherapy program will be applied 2 days a week, 60 minutes a day for 10 weeks and consist of weight bearing on the upper and lower extremities, strengthening, functional stretching exercises, walking training and balance exercises.
Other: Video Game Based Exercise Training — In the Video Game Based Exercise Training program, in addition to the same conventional physiotherapy application for 30 minutes a day, 2 days a week for 10 weeks, 30 minutes of Microsoft Xbox Kinect video games such as reflex ridge and rallyball are used.
  Arms: Video Game Based Exercise Training Group

SUMMARY:
Cerebral palsy (CP) is a non-progressive neurological disorder characterized by a persistent decline in sensory, cognitive or especially gross and fine motor functions during infancy or early childhood. In children with spastic CP, spasticity, muscle weakness, delay in motor development, inadequacy of gross and fine motor skills, selective motor control and functional capacity may be affected. Selective motor control (SMC) is the ability to isolate a muscle or muscle group to perform a specific movement. In children with CP, spasticity directly causes impairment of SMC, as movement patterns governed by flexor or extensor synergies are affected, which inhibits functional movements. Motor dysfunction in CP causes activity limitations and can negatively affect functional capacity. In addition, falls may increase in individuals with CP due to poor balance control, resulting in pain, injury and disability, and may cause individuals to lose confidence in their ability to perform routine activities. Increased fear of falling in individuals with CP may also lead to restriction of activities.It was discussed that the interactive computer game has possible evidence of efficacy allowing to improve gross motor function in individuals with CP. It also appears to have the potential to produce gross motor improvements in terms of strength, balance, coordination and gait for individuals with CP.As a result of our literature review, studies investigating the effect of virtual reality games on gait, balance and coordination in children with CP were observed. However, the effect of virtual reality games on selective motor control has not been sufficiently investigated. The aim of our study, which is planned to eliminate this deficiency in the literature, is to investigate the effect of video game-based exercise training, which provides higher motivation than conventional physical therapy methods, on selective motor control, fear of falling and functional capacity in individuals with CP.

DETAILED DESCRIPTION:
The effect of Virtual Reality Kinect video games, which provide higher motivation than conventional physical therapy methods, on selective motor control, fear of falling and functional capacity will be examined.

The study will include children with spastic CP between the ages of 6-18 years who are attending a Special Education and Rehabilitation Center and who agree to participate in the study. According to the power analysis based on the reference article, it is planned to include 26 people in the study, 13 in the convention physiotherapy group and 13 in the video game-based exercise group.

The families of the children included in the study will be asked to sign an Informed Consent Form and the children will be asked to sign a Child Consent Form for Research Purposes. Demographic data such as gender, age, type of extremity involvement, age at diagnosis will be recorded before the training. The cognitive level of the individuals will be evaluated with the Mini Mental State test, gross motor levels will be classified according to the Gross Motor Function Classification System and hand skills will be classified according to the Hand Skills Classification System. Selective motor control of the upper extremity will be evaluated with the Selective Control of Upper Extremity Evaluation Scale (SCUES) and selective motor control of the lower extremity will be evaluated with the Selective Control of Lower Extremity Evaluation Scale (SCALE). Individuals' balance skills in daily living activities will be evaluated with the Pediatric Balance Scale, fear of falling will be evaluated with the Pediatric Fear of Falling Scale, and functional capacity will be evaluated with the 6-minute walk test.

ELIGIBILITY:
Inclusion Criteria

* Being diagnosed with spastic CP
* Being between the ages of 6-18
* Being at level I, II, III according to MACS
* Being at level I, II, III according to GMFCS
* Scoring 24 points and above on the Mini Mental State Examination
* To have adequate communication skills
* The family agrees to the inclusion of their child in the study
* Child's willingness to participate in the study
* Regular attendance to exercise training within the specified time periods

Exclusion Criteria:

* Any botulinum toxin application and surgical intervention to the lower and upper extremities in the last 6 months
* Serious vision and hearing problems
* Children who have difficulty understanding and following the rules of the game,
* Receiving surgery or botox application to the lower or upper extremity
* Individuals with joint contracture
* Those with pacemakers because they emit radio waves

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Selective Voluntary Motor Control of the Upper Extremities (SCUES) | 10 weeks
  SCUES is a test that evaluates selective motor control of the upper extremity with a score between 0-3. SCUES assesses the shoulder, elbow, forearm, wrist and fingers bilaterally. Motion at each of the five joint levels is graded on a four-point scale: Normal Selective Motor Control (3 points) M3, Mildly Diminished Selective Motor Control (2 points) M2, Moderately, Diminished Selective Motor Control (1 point) M1, No Selective Motor Control (0 points) M0. Higher scores mean a better outcomes.
Selective Control Assessment of the Lower Extremity (SCALE) | 10 weeks
  It is a test that evaluates the selective motor control of the lower extremity with a score between 0 and 2. It evaluates the hip, knee, ankle and toe joints bilaterally.Scoring is graded at each joint as 'Normal' (2 points), 'Impaired' (1 point), or 'Unable' (0 points).Higher scores mean a better outcomes.
Six Minute Walk Test (6MWT) | 10 weeks
  The 6MWT is a simple, submaximal, clinical exercise test that measures the distance walked in 6 minutes under controlled conditions. The 6MWT has been used in children with cerebral palsy (CP) in recent years. In these populations, the 6MWT is considered a measure of overall 'functional status' as 6MWT performance involves the integrated response of multiple body systems.
Pediatric Fear of Falling Questionnaire | 10 weeks
  It is a scale that assesses the fear of falling in activities of daily living in the pediatric population. There are 6 main topics. There are a total of 34 items in which children's fear of falling is questioned during different activities. Participants receive a score between 0 and 68, with higher scores indicating higher fear of falling.

SECONDARY OUTCOMES:
Pediatric Balance Scale (PBS) | 10 weeks
  Assesses children's balance and consist of 14 items. Each item is scored between 0 and 4 points. Low score refers to the poor balance and the high score refers to the good balance.
Gross Motor Classification System (GMFCS) | Baseline
  This is a classification system for children with chronic disability and based on the movements initiated by the child him/herself such as sitting, moving and acting. GMFCS classifies gross motor functions of children with CP in five levels. As the level increases, the level of motor function decreases. Individuals at level 1 have better motor function.
Manual Ability Classification System (MACS) | Baseline
  MACS is a five-level classification system that analyzes the children with CP use their hands while carrying objects in their daily activities.Hand function deteriorates as the level increases. Individuals at level 1 have the best manual ability, while individuals at level 5 have the worst manual ability.
Modified Mini Mental Test (MMMT) | Baseline
  The MMMT adapted for children is used to examine cognitive functions in children from the age of 4 years. The test, which takes 5 to 10 minutes to administer, assesses 5 cognitive areas, including orientation, memory, concentration, language functions and measures of structural ability. The total score on the test reaches a plateau at around 9-10 years of age. In children over 10 years of age, scores below 27 out of a total of 35 points are indicative of mental retardation.

CONTACTS AND LOCATIONS:
Overall Officials: Sezen Tezcan, Principal Investigator — Bolu Abant Izzet Baysal University, Faculty of Health Sciences; Süveybe Yavaş, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No